CLINICAL TRIAL: NCT05662462
Title: ACHIEVE: Successfully Achieving and Maintaining Euglycemia During Pregnancy for Type 2 Diabetes Through Technology and Coaching
Brief Title: Successfully Achieving and Maintaining Euglycemia During Pregnancy for Type 2 Diabetes Through Technology and Coaching
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Kartik K Venkatesh, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022H0399
Record Dates: First submitted 2022-11-22; First posted 2022-12-22 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Pre-Gestational Diabetes; Type2diabetes; Pregnancy in Diabetic; Pregnancy, High Risk
Keywords: mHealth; Pregnancy; Type 2 diabetes; Continuous glucose monitoring; Mobile application; Medicaid; Glycemic control
MeSH Terms: conditions — Pregnancy in Diabetics; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessment of the primary outcome of glycemic control (Hemoglobin A1c <6.5%) will assessed blinded to study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- ACHIEVE Intervention (Active Comparator): The intervention includes a multi-component, including a mobile health (mHealth) application (app), provider dashboard, DEXCOM continuous glucose monitoring (CGM), and care team coaching for medical and social needs. The intervention group will also receive standard of care as described below.
  Interventions: Device: DEXCOM G7 PRO Continuous Glucose Monitor; Device: Patient mHealth app linked to a provider dashboard; Behavioral: Care team coaching for medical and social needs (HUB); Device: Provider dashboard
- Standard of care (No Intervention): Standard of care includes prenatal visits, self-monitored blood glucose, and certified diabetes care and education specialist support.

INTERVENTIONS:
Device: DEXCOM G7 PRO Continuous Glucose Monitor — Participants in the intervention arm will be provided with DEXCOM® G7 PRO CGM sensors and transmitters. The Dexcom G7 CGM system is accurate and safe in pregnant individuals with diabetes. Participants will be taught how to place and remove CGM sensors by a trained research nurse, and will be given sensors to change themselves at home every 10 days. Of note, the DEXCOM® G7 PRO can be applied as a patch on the abdomen, arm, or upper buttocks, is well-tolerated in pregnancy, and does not require calibration. Our mHealth app will allow for wireless synchronization with the CGM sensor so that data are seamlessly reported back to the healthcare team.
  Arms: ACHIEVE Intervention
Device: Patient mHealth app linked to a provider dashboard — The mHealth app is based on our team's prototype intervention developed at our study site. The mHealth app provides diverse functions, including education, reminders, care goals, care pathway recommendations, CGM data and PROs reporting and monitoring, messaging and video conferencing, and a calendar function. Content is based on clinical guidelines for diabetes in pregnancy. Participants will be directed to appropriate resources and online learning to help them navigate the app and its resources. PROs in the mHealth app will be embedded to address health and social needs, and rule-based algorithms will provide tailored care goals, show care pathways, and establish the frequency of elicited PROs.
  Arms: ACHIEVE Intervention
Behavioral: Care team coaching for medical and social needs (HUB) — Participants will be screened at enrollment and throughout the intervention for social needs using a survey adapted from validated instruments, such as the Accountable Health Communities Health-Related Social Needs Screening Tool. The care team will refer participants with affirmative responses to the HUB through the provider dashboard to address social needs (e.g., food insecurity, housing, employment). HUB community health workers will perform comprehensive social needs assessments and connect participants to community resources through "care pathways," a defined action plan addressing patient needs which is recorded and tracked.
  Other Names: Healthcare Collaborative of Greater Columbus Central Ohio Pathways HUB and social needs
  Arms: ACHIEVE Intervention
Device: Provider dashboard — The ACHIEVE intervention will include a bi-directional dashboard that displays information about individuals, including priority care goals and pathways, and recommendations generated via PROMPT. Healthcare team members can access the dashboard embedded within a portal to modify or update information and close the loop on participant tasks. The dashboard will present recommendations for participant goals and pathways provided by the PROMPT algorithms. Providers can use these recommendations or manually select ones for the participant. Providers can sequence goals and pathways by level of complexity. Both the HUB and the healthcare team can perform ongoing assessments of HUB pathway selections and assess recurring needs through the provider dashboard.
  Arms: ACHIEVE Intervention

SUMMARY:
The ACHIEVE RCT will measure the effect of the intervention (mHealth app with CGM, provider dashboard, and care team coaching) compared to current standard care (prenatal visits, self-monitored blood glucose, and certified diabetes care and education specialist) on achieving glycemic control (hemoglobin A1c <6.5% in the third trimester). We hypothesize a 25% absolute increase in the proportion of participants in the intervention group who will meet the target hemoglobin A1c <6.5% in the third trimester compared to the standard care group

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) in pregnancy increases the risk of adverse outcomes for both the mother and infant. Over 1 in 3 infants born to individuals with T2D will experience an adverse outcome, including large for gestational age at birth, preterm birth, birth trauma, neonatal hypoglycemia, and stillbirth. Strict maternal glycemic control throughout pregnancy is key to optimizing perinatal outcomes. This is possible with insulin pharmacotherapy, vigilant glucose monitoring, lifestyle modifications including diet and exercise, and team-based prenatal care. Medicaid-enrolled pregnant individuals with T2D experience non-medical social needs that limit their ability to achieve glycemic control, including lack of reliable transportation to attend prenatal visits, access to resources to engage in diet and exercise changes, and convenient methods to log self-monitored glucose values and adjust insulin dosing.

A multi-faceted provider-patient based approach is needed with proven strategies to improve glycemic control. We propose "ACHIEVE: Successfully achieving and maintaining euglycemia during pregnancy for type 2 diabetes through technology and coaching." Our intervention is multi-component, including a mobile health (mHealth) application (app), provider dashboard, DEXCOM continuous glucose monitoring (CGM), and care team coaching for medical and social needs. This intervention empowers Medicaid-enrolled pregnant individuals with T2D and their healthcare providers to achieve and maintain glycemic control, improve access to care, and provide patient education and support. Each sub-component of the proposed intervention is grounded in Social Cognitive Theory (SCT), and emphasizes on individuals' skills, knowledge and beliefs, and self-efficacy to achieve glycemic control.

We propose four aims: AIM 1: Develop the tailored ACHIEVE mHealth app and provider dashboard for Medicaid-enrolled pregnant individuals with T2D and their healthcare team through active stakeholder engagement; AIM 2: Conduct an RCT and measure the effect of the intervention (mHealth app with CGM, provider dashboard, and care team coaching) compared to current standard care (prenatal visits, self-monitored blood glucose, and certified diabetes care and education specialist) on achieving glycemic control (hemoglobin A1c <6.5% in the third trimester). We hypothesize a 25% absolute increase in the proportion of participants in the intervention group who will meet the target hemoglobin A1c <6.5% in the third trimester compared to the standard care group; and AIM 3: Identify multi-level patient and provider barriers and facilitators to satisfaction, engagement, and use of the intervention and its subcomponents. AIM 4: Examine postpartum (i.e. 6-12 months after delivery) diabetes and reproductive health outcomes in both intervention and standard care arms.

ELIGIBILITY:
Inclusion Criteria:

1. pregnant individuals age ≥18 years;
2. ≤20 weeks of gestation (specifically, <20+6 weeks);
3. diagnosis of pregestational T2D and A1c ≥6.5% at the time of study enrollment;
4. Medicaid insurance;
5. English or Spanish speaking;
6. cognitively able to complete the study requirements;
7. consent to all study activities;
8. accessible for participation in study activities;
9. use a smartphone with internet access;

Participants must also consent to the study team abstracting information from their electronic health records (EHRs), using CGM for glucose monitoring if randomized to the intervention group, tracking the participants' clinic, hospital, and emergency room visits during the study period, as well as tracking the number of times the participants use the ACHIEVE mobile health (mHealth) application (app), including what activities are used in the mobile application (e.g., recording blood glucose, scheduling appointments, messaging their healthcare providers, accessing educational resources).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is restricted to pregnant individuals.
Enrollment: 124 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
The primary clinical outcome is the proportion of participants with an A1c <6.5% in the third trimester before delivery | From ≤20 weeks of gestation to delivery, an average of 5 months
  A1c is a blood test that represents the average glucose over the previous three months. Our outcome threshold is slightly higher than the target of <6.0 recently recommended by ADA because: 1) our target population of pregnant individuals includes those with poor glycemic control at enrollment, 2) an aggressive target <6% can result in frequent episodes of hypoglycemia, of particular concern for participants in the standard care arm without CGM, and 3) the frequency of adverse neonatal outcomes are similar with third trimester A1c 6-6.4% vs. <6%. A1c will be assessed once per trimester, consistent with ADA and ACOG guidelines for T2D management in pregnancy, and at delivery. For participants with >1 value in the third trimester, the value closest to delivery will be used. A standard assay will be used for HbA1c. We will evaluate HbA1c as an absolute percentage of total hemoglobin using reference standards per the Diabetes Control and Complications Trial Reference Method.

SECONDARY OUTCOMES:
Large for gestational age at birth | At birth
  Birthweight >90% for gestational age using a 2017 NCHS reference standard
Neonatal hypoglycemia | 48 hours of delivery
  Any blood glucose <30 mg/dL within 48 hours of delivery
NICU admission | Delivery admission
  NICU admission for any indication
Preterm birth <37 weeks | At birth
Respiratory distress syndrome | Delivery admission
Percentage of time-in-range (TIR) | Across pregnancy from randomization to delivery, which is approximately from 12 weeks to 38 weeks gestation or 26 weeks total
  Among participants in the intervention arm, we will assess CGM measures of glycemic control. The target range will be between 63 to 140 mg/dL, consistent with the CONCEPTT CGM trial in pregnant individuals with T1D, emerging data in pregnancy, and expert opinion. We will assess TIR as both a continuous and dichotomous measure (≥85%).
Mean CGM glucose levels during the day and night | Across pregnancy from randomization to delivery, which is approximately from 12 weeks to 38 weeks gestation or 26 weeks total
  Among participants in the intervention arm, we will assess CGM measures of glycemic control.
Time spent above and below target range | Across pregnancy from randomization to delivery, which is approximately from 12 weeks to 38 weeks gestation or 26 weeks total
  Among participants in the intervention arm, we will assess CGM measures of glycemic control.
Low and high blood glucose indices | Across pregnancy from randomization to delivery, which is approximately from 12 weeks to 38 weeks gestation or 26 weeks total
  Among participants in the intervention arm, we will assess CGM measures of glycemic control.
Patient activation measure (PAM) | Once per trimester (~12 weeks, 24 weeks, and 36 weeks)
  These outcomes will be measured by survey to capture knowledge, skill, and confidence to manage one's health and health care 13-items, continuous scale measures from 0 to 100. This is a PRO.
Patient intervention tool technology engagement | Across pregnancy from randomization to delivery, which is approximately from 12 weeks to 38 weeks gestation or 26 weeks total
  Patient intervention tool technology engagement data will be collected through Log files and will be measured as the number of sessions a participant had with the tool (total and average use for tool and specific functions).
The Accountable Health Communities. Health-Related Social Needs Screening Tool | Across pregnancy from randomization to delivery, which is approximately from 12 weeks to 38 weeks gestation or 26 weeks total
  Provider dashboard and HUB data (for intervention group) and EHR referral and chart notes by licensed social worker (standard of care group).
Blood glucose levels | Across pregnancy from randomization to delivery, which is approximately from 12 weeks to 38 weeks gestation or 26 weeks total
  EHR data and mHealth app (CGM)(for the intervention group) and self-monitored blood glucose (for standard of care group)
Diabetes Knowledge Questionnaire (DKQ) | Once per trimester (~12 weeks, 24 weeks, and 36 weeks)
  Measured through Patient's Diabetes Knowledge Questionnaire. This is a PRO. 24 item scale, continuous measure.
Morisky Medication Adherence Scale (MMAS-8) | Across pregnancy from randomization to delivery, which is approximately from 12 weeks to 38 weeks gestation or 26 weeks total
  Adherence will be measured through Medication Adherence Scale. This is a PRO
Health care utilization | Across pregnancy from randomization to delivery, which is approximately from 12 weeks to 38 weeks gestation or 26 weeks total
  Scheduled prenatal clinic visits, hospitalizations, emergency department visits, obstetric triage visits, and unscheduled clinic visits through EHR. Data will be collected from the electronic health record and patient survey.
Short Assessment of Health Literacy-Spanish and English (SAHL-S&E) | Once per trimester (~12 weeks, 24 weeks, and 36 weeks)
  Health literacy will be measured through eHealth literacy scale and Health literacy scale. This is a PRO. A score between 0 and 14 suggests the examinee has low health literacy.
eHealth literacy scale (eHEALS) | Once per trimester (~12 weeks, 24 weeks, and 36 weeks)
  8-item measure of eHealth literacy.
Comprehension of education material | 3 times in the first six weeks and then monthly during study participation, which is approximately from 12 weeks to 38 weeks gestation or 26 weeks total.
  Comprehension of education material will be measured through Self-developed survey. This is a PRO.
Diabetes Distress Scale (DDS) | Once per trimester (~12 weeks, 24 weeks, and 36 weeks)
  Diabetes Distress will be measured through the Diabetes Distress Scale. This is a PRO. The DDS is a self-report survey that has 17 items.
Self-efficacy for Diabetes | Across pregnancy from randomization to delivery, which is approximately from 12 weeks to 38 weeks gestation or 26 weeks total.
  Self-efficacy will be measured through the Diabetes Management Self-Efficacy Scale. This is a PRO. Continuous measure or mean score of 8 items.
Doctor-Patient Communication Scale | Across pregnancy from randomization to delivery, which is approximately from 12 weeks to 38 weeks gestation or 26 weeks total
  The questionnaire contains 15 items with 4 possible answers: no, possibly no, possibly yes, and yes, rated according to a Likert-type scale (1 to 4 points), with score of 4 being the best possible response.

CONTACTS AND LOCATIONS:
Overall Officials: Naleef Fareed, PhD, MBA, Principal Investigator — Ohio State University; Joshua J Joseph, MD, Principal Investigator — Ohio State University; Kartik K Venkatesh, MD, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center OB/GYN Maternal and Fetal Medicine, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Venkatesh KK, Joseph JJ, Swoboda C, Strouse R, Hoseus J, Baker C, Summerfield T, Bartholomew A, Buccilla L, Pan X, Sieck C, McAlearney AS, Huerta TR, Fareed N. Multicomponent provider-patient intervention to improve glycaemic control in Medicaid-insured pregnant individuals with type 2 diabetes: clinical trial protocol for the ACHIEVE study. BMJ Open. 2023 May 10;13(5):e074657. doi: 10.1136/bmjopen-2023-074657. PMID 37164461